CLINICAL TRIAL: NCT04321876
Title: Evaluation of a Collaborative Behavioral Health Program Implementation in Primary Care
Acronym: WBCBHP
Status: Active, not recruiting | Type: Observational
Sponsor: Northwestern University (Other)
Collaborators: Northwestern Medicine (Other)
Responsible Party: Principal Investigator, Allison Carroll, Assistant Professor, Northwestern University
Other Study IDs: STU00208338
Record Dates: First submitted 2020-03-23; First posted 2020-03-25 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-04

CONDITIONS: Depression
Keywords: primary care; collaborative care model; implementation
MeSH Terms: conditions — Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (11):
- NMG IM 211 E Chicago Ave
  Interventions: Behavioral: Collaborative Behavioral Health Program
- NMG IM ARKES
  Interventions: Behavioral: Collaborative Behavioral Health Program
- NMG IM 1460 N Halsted St
  Interventions: Behavioral: Collaborative Behavioral Health Program
- NMG IM 201 E Huron St
  Interventions: Behavioral: Collaborative Behavioral Health Program
- NMG Integrative Medicine 150 E Huron St
  Interventions: Behavioral: Collaborative Behavioral Health Program
- NMG IM 1776 N Milwaukee Ave
  Interventions: Behavioral: Collaborative Behavioral Health Program
- NMG IM 20 S Clark St
  Interventions: Behavioral: Collaborative Behavioral Health Program
- NMG IM FM 1704 Maple Ave
  Interventions: Behavioral: Collaborative Behavioral Health Program
- NMG IM 259 E Erie St
  Interventions: Behavioral: Collaborative Behavioral Health Program
- NMG IM 1135 S Delano Ct
  Interventions: Behavioral: Collaborative Behavioral Health Program
- NMG IM 1333 W Belmont Ave
  Interventions: Behavioral: Collaborative Behavioral Health Program

INTERVENTIONS:
Behavioral: Collaborative Behavioral Health Program — Collaborative care is the delivery of mental health care through a proactive collaboration of primary care providers, behavioral care managers based in primary care practices, and psychiatrists who provide supervision to the behavioral care managers and consultation to the primary care providers.

SUMMARY:
This study will give researchers the opportunity to evaluate implementation of the Collaborative Behavioral Health Program (CBHP), based on the collaborative care model for depression, which aims to improve practice for physicians and staff; improve care for patients; and improve clinic operations through a model that allows for more efficient identification and referral for care for depression.

DETAILED DESCRIPTION:
This study used a hybrid Type 2 effectiveness-implementation design of a randomized roll-out trial of the Collaborative Care Model for depression (CoCM) in 11 primary care practices in a large healthcare system affiliated with an academic medical center. The Collaborative Behavioral Health Program (CBHP) is supported by leaders in the healthcare system and the primary care steering committee as a means of improving access to effective mental health services. Implementation strategies including hiring and training the necessary staff for CoCM, audit and feedback procedures, and health information technologies to assist with billing and the patient registry, will be provided for all practices. Using a sequential mixed methods measurement approach, we will assess key stakeholders' perspectives of CBHP roll-out, focused on barriers and facilitators of implementation and sustainability. The Stages of Implementation tool will be used to measure the speed and quantity of implementation activities completed across the stages of implementation preparation, implementation, and sustainment over a 30-month period for each practice. Effectiveness of CBHP for patient-level outcomes will be conducted on depressive symptoms, graduation rates for CBHP, and spillover effects on chronic health conditions.

With its focus on implementation processes and strategies, this study will elucidate the critical drivers of CoCM implementation that are understudied for a program with such a robust evidence base. This study will also be among the first to conduct economic analyses on a fee-for-service model with the new billing codes for CoCM and can inform ways to improve implementation efficiency with our optimization approach to successive practices in the roll-out design. Changes to the protocol and current status of the study are also discussed.

ELIGIBILITY:
Inclusion Criteria:

• PHQ-9 score > 10

Exclusion Criteria:

* Current suicidality
* Bipolar disorder
* Substance abuse disorder
* Psychosis
* Other severe mental health condition

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients attending primary care appointments within the Northwestern Medicine health system's central region.
Sampling Method: Non-Probability Sample
Enrollment: 778 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Impact of implementation strategies on the speed of CBHP implementation (time, in days) | 2 years
  Trends in the rate at which CBHP is implemented over successive practices, as assessed by the Universal Stages of Implementation Completion (USIC)
Impact of implementation strategies on the quantity of CBHP implementation (number of CBHP participants) | 2 years
  Trends in the number of CBHP participants over successive practices, as assessed by CBHP referrals, engagement, and treatment completion derived from the electronic health record
Acceptability of CBHP | 2 years
  Self-report of key stakeholders and CBHP utilization (referral, engagement, completion)
Effectiveness of CBHP on depressive symptoms (PHQ-9 scores) | 2 years
  Pre- and post-treatment self-reported depressive symptoms (PHQ-9 scores), anti-depressant medication prescriptions and adherence, treatment engagement, psychiatry referrals
Effectiveness of CBHP on behavioral health service utilization (antidepressant medication prescription, CBHP treatment engagement, and external referrals for behavioral health) | 2 years
  Proportion of patients who are eligible for CBHP who receive behavioral health services, including anti-depressant medication prescriptions, CBHP treatment sessions, and/or external referrals for behavioral health (e.g., psychiatry)

CONTACTS AND LOCATIONS:
Locations (1):
- Northwestern Medicine, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Smith JD, Hasan M. Quantitative approaches for the evaluation of implementation research studies. Psychiatry Res. 2020 Jan;283:112521. doi: 10.1016/j.psychres.2019.112521. Epub 2019 Aug 17. PMID 31473029
- [Derived] Kordon A, Carroll AJ, Fu E, Rosenthal LJ, Rado JT, Jordan N, Brown CH, Smith JD. Multilevel perspectives on the implementation of the collaborative care model for depression and anxiety in primary care. BMC Psychiatry. 2024 Jul 22;24(1):519. doi: 10.1186/s12888-024-05930-w. PMID 39039458